CLINICAL TRIAL: NCT05468684
Title: The Course and Neuroplasticity in Neck Pain-Associated Disorders and Whiplash-Associated Disorders in the General Population: A One Year Prospective Observational Cohort Study PROCO-Neck
Brief Title: PROCO Neck: The Course and Neuroplasticity in Neck Pain-Associated Disorders and Whiplash-Associated Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: University of applied sciences (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 32003B_205101/1
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Neck Pain; Whiplash; Pain, Acute; Psychosocial Functioning; Activity, Motor; Alteration of Cognitive Function; Pain, Chronic; Pain Catastrophizing; Overactivity; Behavior
MeSH Terms: conditions — Neck Pain; Whiplash Injuries; Acute Pain; Motor Activity; Chronic Pain; Spasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neck Pain-Associated Disorders: neck pain without an acceleration-deceleration mechanism
  Interventions: Other: no intervention
- Whiplash-Associated Disorders: neck pain resulting from a traumatic acceleration-deceleration mechanism and classified as WAD Grade I-III on the modified Quebec Task Force Scale
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there are no interventions planned, we observe the patients in a cohort study which is named inception cohort study because we test participants before the condition develops.

SUMMARY:
Neck pain-associated disorders (NAD) and whiplash-associated disorders (WAD) are major health problems. NAD has a lifetime prevalence of 54%. Although the majority of patients recovers within the first three months, a minority develops persistent pain. WAD, in contrast, is reported less frequently, but patients are often suffering more badly. Patients with chronic symptoms represent a considerable burden in terms of pain, suffering, health care needs, and social costs. Findings on the natural course of NAD and WAD reflect the necessity to identify factors besides pain related to the persistence of symptoms. First, alterations of input and processing of multiple sensory modalities causing movement control impairment can result in persistent symptoms and affect the quality of life. Besides, findings of psychosocial factors predictive of pain outcomes support the growing body of research proposing a bidirectional relationship between somatic and psychosocial variables. In particular, there is a pressing need to investigate pain-related activity patterns, besides fear-avoidance behavior in NAD and WAD. Maladaptive activity pattern have an impact on on pain and disability in the long-term prognosis. Mt important, given the high prevalence of NAD and WAD, the cortical representation of the cervical spine has not yet been investigated and, reports on neuroplasticity remain scarce. These shortcomings should be addressed to provide evidence for the temporal aspect of neuroplasticity and its involvement in pain persistence.

Hypotheses:

We hypothesize I. that impaired sensorimotor abilities, mental health at baseline increase pain intensity and disability during measurement.

II. that maladaptive pain-related activity patterns avoidance and overactivity at baseline are prognostic factors for pain persistence and disability.

III. that the WAD cohort shows more depression, anxiety and stress compared to the NAD cohort.

DETAILED DESCRIPTION:
The proposed project comprises two parts. The prospective study will assess clinical and cognitive behavioral data at four time points (1-3-6-12 months) after the onset of pain. Part I investigates sensorimotor functioning and cognitive-behavioral variables in NAD and WAD, using state-of-the-art clinical assessments and questionnaires presented in an online survey. Part II explores for the first time the representation of the cervical spine in a control group and, subsequently investigates neuroplastic changes in sensorimotor networks. The association of clinical testing, questionnaire, and neuroimaging data may act as indicative factors for the development of persistent symptoms in NAD and WAD, respectively protective mechanisms in a remission of symptoms. We aim to gain insights into the time-related process of NAD and WAD - its similarities and differences - resulting from the changes in sensory processing, movement performance, and their interaction with cognitive-behavioral factors. The prospective approach might shed light on time dependent processes during the transition from acute to a persistent pain state. The proposed research is user-driven and has the potential to be translated into a target group-oriented assessment and treatment of NAD and WAD by a variety of health care professionals.

Primary Aims:

I. To observe functional, clinical, and psychosocial variables by using clinical tests and online surveys for 12 months in acute NAD and WAD cohorts in the working-age population.

II. To investigate the course and stability of pain-related activity patterns III. Compare functional, clinical, and psychosocial variables between NAD and WAD cohorts.

Experimental time points:

The proposed study design is an observational longitudinal cohort study investigating functional, clinical, and psychosocial factors in NAD and WAD patients over one year. The study protocol comprises four-measurement points at 1-3-6-12 months after the onset of pain.

Recruitment process:

In a simple random sampling, patients will be recruited from local physiotherapists and general practitioners (GP) when presenting with NAD and WAD. Furthermore, information flyers and posters will be distributed in various medical associations (hospitals, massage practice). Then, we will use e-mail distribution within affiliates of the University of Zurich and the ZHAW. Finally, we will call on different social media channels like Facebook and Twitter.

Psychometric instruments We will collect demographic and questionnaire data using the online survey tool REDCap (Research Electronic Data Capture, https://projectredcap.org/software/), widely used in the academic research community for flexible and robust data collection. The application of online surveys reduces costs and time, including automated checks for plausibility and completeness. Participants are more diverse demographically than the paper-and-pencil method, and both ways revealed similar results.

ELIGIBILITY:
Inclusion Criteria:

* NAD cohort; neck pain without an acceleration-deceleration mechanism, inclusion < 1 month since onset of pain
* WAD cohort; neck pain resulting from a traumatic acceleration-deceleration mechanism and classified as WAD Grade I-III on the modified Quebec Task Force Scale98, inclusion < 1 month since onset of pain
* In recurrence, no pain in the previous three months
* Age between 18 and 65 years at baseline
* Ability to read, write, and understand German for completing the questionnaires.

Exclusion Criteria:

* For both cohorts; a clinically relevant anatomical anomaly in the cervical spine (e.g., carcinoma), spine surgery; peripheral or central neurological illness, pregnancy, or women who gave birth in the last year (to avoid the confounding effects of pregnancy-related NAD)
* For the WAD cohort, WAD Grade IV on the modified Quebec Task Force Scale (Fracture of dislocation), patients who lost consciousness due to the traumatic event and post-traumatic amnesia to exclude mild traumatic brain injury.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with acute NAD or acute WAD, 18-65 years old with the ability to read, write, and understand German.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 1 year
  Numeric Rating Scale (NRS). The NRS is a single 11- point numeric scale ranging from 0 to 10, with 0 representing "no pain" and 10 representing "worst pain you can imagine".
Disability | 1 year
  German version of the Neck Disability Index (NDI-G). The self-administered questionnaire consists of 10 items referring to various activities (personal care, lifting, driving, work, sleeping, concentration, reading, recreation) and pain (pain intensity, headache) with 6 possible answers per item. Each item is scored from 0 (no pain and no functional limitation) to 5 (worst pain and maximal limitation) points resulting in a minimal score of 0 points (no disability) to a maximum possible score of 50 points (totally disabled)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hotz-Boendermaker, Principal Investigator — University of applied sciences
Locations (1):
- Zurich University of Applied Sciences: School of Health Sciences, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morf R, Kernwein C, Jaeger J, Reicherzer L, Degenfellner J, Hotz-Boendermaker S. Prognostic value of activity patterns and stress measures for persistent pain and disability in acute neck pain: a 3-month follow-up study. Front Pain Res (Lausanne). 2025 Nov 13;6:1686389. doi: 10.3389/fpain.2025.1686389. eCollection 2025. PMID 41322119